CLINICAL TRIAL: NCT02773563
Title: Role of CO2 Insufflation vs. Air Insufflation for Endoscopic Ultrasound: a Prospective Observational Study
Brief Title: CO2 vs. Air Insufflation for Endoscopic Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pietro Fusaroli, Associate professor, University of Bologna
Other Study IDs: 2016/001
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Lesion; Gastrointestinal; Liver, Biliary, Pancreas and Gastrointestinal Disease, Nos
MeSH Terms: conditions — Gastrointestinal Diseases; Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EUS with CO2 insufflation: Patients undergoing EUS with CO2 insufflation
  Interventions: Other: EUS with CO2 insufflation
- EUS with air insufflation: Patients undergoing EUS with air insufflation
  Interventions: Other: EUS with air insufflation

INTERVENTIONS:
Other: EUS with air insufflation — Diagnostic procedure using an echoendoscope for the study of pancreaticobiliary or gastrointestinal diseases using air insufflation
  Groups: EUS with air insufflation
Other: EUS with CO2 insufflation — Diagnostic procedure using an echoendoscope for the study of pancreaticobiliary or gastrointestinal diseases using CO2 insufflation
  Groups: EUS with CO2 insufflation

SUMMARY:
The insufflation of air in the viscera is indispensable during endoscopy. However, the distension of the bowel that follows is often the cause of abdominal discomfort.

Carbon dioxide (CO2) has been widely used for insufflation in endoscopy. CO2 insufflation is demonstrated in the literature to cause lower abdominal discomfort as it is quickly reabsorbed by the body.

Endoscopic ultrasonography (EUS) is a method in which you associate the endoscopic view and the ultrasound vision obtained from the inside of the viscera.

The diagnostic accuracy of EUS is undermined by the visual artifacts caused by the presence of air between the probe and the organ to be studied.

Although the use of CO2 is already widely applied by many endoscopists, there are no studies to date concerning the use of CO2 during EUS from the point of view of the abdominal discomfort related to the procedure and/or the quality of the images obtained.

The main purpose of the study is to assess whether the insufflation of CO2 results in a reduction of discomfort of the patients undergoing EUS. The study design is observational because no randomization or other interventions are planned; participants will be assigned to either air or CO2 insufflation according to the endoscopic room equipment (one room is equipped with CO2 insufflation while another endoscopic room is equipped just with air insufflation) and the results of the two groups will be compared. Among the secondary goals the investigators want to evaluate whether insufflation of CO2 is associated with a reduction in the dose required for patients sedation. Finally, the investigators want to clarify whether the use of CO2 is able to produce less visual artifacts than air and thus improve the quality of EUS images.

DETAILED DESCRIPTION:
The insufflation of air in the viscera during endoscopy is indispensable in order to allow the advancement of endoscopic probe, to visualize the mucosa and to avoid injury to the gastrointestinal wall. However, the distension of the bowel that follows is often the cause of abdominal discomfort since the air blown appears to be slightly absorbable and therefore it needs a long time to be expelled.

Carbon dioxide (CO2) is a gas that has already been widely used for insufflation in endoscopy. CO2 insufflation is demonstrated in the literature to cause lower abdominal discomfort as it is quickly reabsorbed by the body. This gas is at the same time devoid of side effects.

Studies in the literature focus mainly on the intensity of abdominal discomfort after the insufflation of CO2 vs. air while performing colonoscopy, endoscopic retrograde cholangiopancreatography (ERCP) and enteroscopy.

Endoscopic ultrasonography (EUS) is a method in which you associate the endoscopic view and the ultrasound vision obtained from the inside of the viscera. The main indications to EUS are represented by the study of the biliary pancreatic diseases, the staging of the digestive tract tumors and the differential diagnosis of submucosal tumors.

The diagnostic accuracy of EUS is undermined by the visual artifacts caused by the presence of air between the probe and the organ to be studied; during the procedure the endoscopist must ensure, by means of repeated suctions, that the least possible amount of air is present inside the viscera.

Although the use of CO2 is already widely applied by many endoscopists, there are no studies to date concerning the use of CO2 during EUS from the point of view of the abdominal discomfort related to the procedure and/or the quality of the images obtained.

At the moment, with regard to EUS, there are no recommendations regarding the use of a gas rather than the other; the choice is in fact at the discretion of the operator and also it depends on the availability in the individual endoscopic units of the instrumentation for CO2 insufflation.

At Our Endoscopic Unit, CO2 or air insufflation is decided upon the availability of the equipment in the endoscopic room; in particular, in Suite 1, patients receive air insufflation and in Suite 2 they receive CO2 insufflation. The assignment into one or the other endoscopic room is purely casual according to scheduling the next free available slot.

The main purpose of the study is to assess whether there is any difference between CO2 and air insufflation in inducing discomfort of the patients undergoing EUS. The study design is observational because no randomization or other intervention modifications are planned; participants will be assigned to either air or CO2 insufflation according to the endoscopic room equipment (one room is equipped with CO2 insufflation while another endoscopic room is equipped just with air insufflation) and the results of the two groups will be compared. Among the secondary goals the investigators want to evaluate whether insufflation of CO2 is associated with a reduction in the dose required for patients sedation. Finally, the investigators want to clarify whether the use of CO2 is able to produce less visual artifacts than air and thus improve the quality of EUS images.

ELIGIBILITY:
Inclusion Criteria:

• Consecutive patients referred for EUS

Exclusion Criteria:

* Age <18
* Pregnancy
* Unwillingness to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indications for undergoing EUS (in general they are represented by patients with pancreaticobiliary or gastrointestinal diseases)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Abdominal discomfort | through study completion, an average of 1 year
  Self reported pain measurement after endoscopic ultrasound assessed with a Visual Analog Scale (VAS 0-10)

SECONDARY OUTCOMES:
Dose of sedation | through study completion, an average of 1 year
  Measured by the physician after endoscopic ultrasound
Quality of EUS images | through study completion, an average of 1 year
  Evaluation of the quality of EUS images by several physicians

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Fusaroli, MD, Principal Investigator — Department of Medical and Surgical Sciences, GI Unit, University of Bologna/Hospital of Imola, Imola, Italy
Locations (1):
- Gastrointestinal Unit, University of Bologna/Hospital of Imola, Imola (BO), Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Hu B. The role of carbon dioxide insufflation in colonoscopy: a systematic review and meta-analysis. Endoscopy. 2012 Feb;44(2):128-36. doi: 10.1055/s-0031-1291487. Epub 2012 Jan 23. PMID 22271023
- [Background] Bretthauer M, Lynge AB, Thiis-Evensen E, Hoff G, Fausa O, Aabakken L. Carbon dioxide insufflation in colonoscopy: safe and effective in sedated patients. Endoscopy. 2005 Aug;37(8):706-9. doi: 10.1055/s-2005-870154. PMID 16032487
- [Background] Li X, Zhao YJ, Dai J, Li XB, Xue HB, Zhang Y, Xiong GS, Ohtsuka K, Gao YJ, Liu Q, Song Y, Fang JY, Ge ZZ. Carbon dioxide insufflation improves the intubation depth and total enteroscopy rate in single-balloon enteroscopy: a randomised, controlled, double-blind trial. Gut. 2014 Oct;63(10):1560-5. doi: 10.1136/gutjnl-2013-306069. Epub 2014 Mar 13. PMID 24626435